CLINICAL TRIAL: NCT03829826
Title: Efficacy and Mechanism of Action of SCIg in Patients With Stiff Person Syndrome
Brief Title: Efficacy and Mechanism of Action of SCIg in Patients With Stiff Person Syndrome (SPS)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 18P.420
Record Dates: First submitted 2019-01-07; First posted 2019-02-04 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Stiff-Person Syndrome
MeSH Terms: conditions — Stiff-Person Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood drawn for humoral (immunological) studies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Patients receiving IVIg: Patients are currently receiving IVIg regularly for at least every 6 weeks and exhibit a favorable response will be recruited into the study (11 patients). They will be observed for 12 weeks under their existing IVIg regimen and will undergo measurements of their impairment using the previously validated Stiffness and Sensitivity scales and quality of life questionnaire (QoL) at weeks 0, 4, 8, 12. At week 12, prior to the first SCIg infusion, blood will be drawn for humoral (immunological) studies. One week following the last dose of IVIg (at week 13), the participants will be started on SCIg at a total dose equivalent to the monthly dose of IVIg they have been receiving.
  Interventions: Biological: HyQvia
- de novo SCIg patients/IVIg-Naive Group: This other arm of the trial will include 11 patients naïve to IVIg who do not receive other immunotherapies while being symptomatic. These patients after a 12-week observation period will start directly on SCIg drug (HYQVIA), following the same schedule as described above for the previous group.
  Interventions: Biological: HyQvia

INTERVENTIONS:
Biological: HyQvia — Immune Globulin Infusion 10% (Human) with Recombinant Human Hyaluronidase

SUMMARY:
This is a pilot, proof-of concept investigator-initiated trial planned for 22 patients with the diagnosis of Stiff Person Syndrome (SPS). The study will compare efficacy of treatment using subcutaneous immunoglobulin therapy (SCIg) compared to intravenous immunoglobulin (IVIg) therapy. The majority of IVIg naïve subjects (those not already receiving IVIg) are typically managed with non-immunotherapy mostly Gamma Aminobutyric Acid (GABA) -enhancing drugs such as Baclofen or Diazepam.

DETAILED DESCRIPTION:
Study Design:This is a proof of concept observational prospective, open label, study on the safety, efficacy and convenience of treatment with SCIg study of 22 patients at Thomas Jefferson University Hospital. Two cohorts of patients within the total of 22 will be included; half of them (11 patients) currently receiving and responding to IVIg and the other half starting de novo on SCIg. Patients diagnosed with SPS according to defined sets of symptoms will be eligible to enroll.

The primary clinical outcome will be based on clinical efficacy measures, as used before for the IVIg trial, based on changes in the Stiffness Index and Heightened Sensitivity scores, using the validated scales that the investigators have had previously utilized and validated (Dalakas et al 2001; see attached at the end of the protocol). These same measurements will be applied while on IVIg (weeks 0, 4, 8, 12) and will be compared to the measurements obtained during SCIg (weeks 16, 20, 24, 28). The secondary outcome will be Quality of Life (QoL) responses and patient preference for each treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged >18 years
* Diagnosis of SPS based on standard criteria
* IVIg Group: Receiving the equivalent of 1-2 g/kg IVIg every 4 weeks with dependence* on IVIg to maintain clinical response *Dependence is clinically determined either by symptomatic worsening of condition at the end of the inter-dose interval or by worsening after dose reduction or discontinuation within the previous 3 months.
* IVIg-Naïve Group: Patients with symptomatic SPS and never treated with IVIg (IVIg-naïve group), poorly controlled with standard therapy

Exclusion Criteria:

* Pregnancy, planned pregnancy, breast-feeding or unwillingness to practice contraception
* Severe concurrent medical conditions, which would prevent treatment or assessment, including significant hematological, renal or liver dysfunction or malignancies
* Initiation of immunomodulatory treatment other than IVIg in the past 3 months
* Participation in a trial of an investigational medicinal product in the past 12 weeks
* Presence of any medical condition, which in the opinion of the investigator might interfere with performance or interpretation of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Yes No Individuals with impaired decision-making capacity X Women of reproductive potential X Pregnant women/fetuses/neonates X Men of reproductive potential X Minorities X Prisoners X Economically or educationally disadvantaged persons X Students/employees X
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
A >50% change from baseline on the Stiffness Index scores ( scale from 0-6; each item adds one) after 12 weeks of treatment. | 24 MONTHS
  Proving that SCIg is as effective as IVIg on this clinical measure will be important for the patients who may have another treatment option avoiding the systemic side effects of IVIg
A >50% change from baseline on the Heightened Sensitivity scores (scales from 1-7, each item adds one) after 12 weeks of treatment. | 24 months
  Proving that SCIg is as effective as IVIg on this clinical measure will be important for the patients who may have another treatment option avoiding the systemic side effects of IVIg

SECONDARY OUTCOMES:
A meaningful change on Quality of Life (QoL) measures after 12 weeks of SCIg based on 6 sets of QoL Questionnaires (mobility, self-care, usual activities, pain, anxiety/depression, health state) | 24 MONTHS
  Proving that SCIg affects Quality of life, as IVIg does, will be important for the patients who may have another treatment option avoiding the systemic side effects of IVIg
If SCIg reduces the anti-GAD antibody titers measured in the patient's blood samples by more than 30% | 24 MONTHS
  An effect on the circulating anti-Glutamic Acid Decarboxylase (GAD) antibodies will elucidate the mechanism of action of SCIg and any correlation between efficacy and antibody titers
If >50% of patients prefer either SCIg or IVIg after 12 weeks of treatment based on a YES/NO questionnaire . | 24 MONTHS
  Proving patients' preference is important because SCIg is self-administered at home and more convenient, without the need for hospitalizations.